CLINICAL TRIAL: NCT02651987
Title: Efficacy and Safety of Lanreotide Autogel® 120 mg Administered Every 14 Days in Well Differentiated, Metastatic or Locally Advanced, Unresectable Pancreatic or Midgut Neuroendocrine Tumours Having Progressed Radiologically While Previously Treated With Lanreotide Autogel® 120 mg Administered Every 28 Days
Brief Title: Efficacy and Safety Study in Pancreatic or Midgut Neuroendocrine Tumours Having Progressed Radiologically While Previously Treated With Lanreotide Autogel® 120 mg
Acronym: CLARINET FORTE
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Ipsen (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 8-79-52030-326; 2014-005607-24 (EudraCT Number)
Record Dates: First submitted 2015-12-11; First posted 2016-01-11 (Estimated); Results first posted 2020-12-30 (Actual); Last update posted 2022-10-03 (Actual); Status verified 2022-09

CONDITIONS: Pancreatic Tumours; Midgut Neuroendocrine Tumours

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Lanreotide Autogel® (Experimental): One subcutaneous (SC) injection of lanreotide Autogel® 120mg every 14 days until disease progression or death or unacceptable toxicity or tolerability.
  Interventions: Drug: Lanreotide autogel 120 mg

INTERVENTIONS:
Drug: Lanreotide autogel 120 mg

SUMMARY:
This study aims to explore the efficacy and safety of lanreotide Autogel® 120 mg administered every 14 days in subjects with grade 1 or 2, metastatic or locally advanced, unresectable pancreatic or intestinal neuroendocrine tumours (NETs) once they have progressed on the standard dose of lanreotide Autogel® 120 mg every 28 days.

ELIGIBILITY:
Inclusion Criteria:

* Histopathologically confirmed, grade 1 or 2, metastatic or locally advanced, unresectable pNET (pNET cohort) or midgut NET (midgut cohort) with or without hormone related syndromes, with a proliferation index (Ki67) ≤20%.
* Positive somatostatin receptors type 2
* Progression as assessed by an independent central reviewer according to RECIST v1.0 while receiving first line treatment with lanreotide Autogel® at a standard dose of 120 mg every 28 days for at least 24 weeks

Exclusion Criteria:

* Grade 3 or rapidly progressive (within 12 weeks) NET
* Any NET other than pancreatic and midgut
* Previous treatment with any antitumour agent for NET other than lanreotide Autogel® 120 mg every 28 days. Exception made of prior treatment with Octreotide at standard dose stopped for other reason than disease progression.
* Symptomatic gallbladder lithiasis at screening echography or history of cholelithiasis with no cholecystectomy since then.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 99 (Actual)
Dates: Start 2015-12-15 (Actual); Primary Completion 2019-10-16 (Actual); Study Completion 2019-10-24 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ipsen Medical Director, Study Director — Ipsen
Locations (32):
- Belgium (4):
  - Erasme Hospital, Brussels
  - Cliniques Unversitaires Saint Luc, Brussels
  - Antwerp University Hospital, Edegem
  - UZ Leuven, Leuven
- Denmark (2):
  - Aarhus University Hospital, Aarhus
  - Rigshospitalet, Copenhagen
- France (4):
  - Hôpital Beaujon, Clichy
  - Hôpital Edouard Herriot, Lyon
  - Institut Paoli Calmette, Marseille
  - Institut Gustave Roussy, Villejuif
- Germany (3):
  - Charité - CVK, Berlin
  - Universitätsklinikum Erlangen, Erlangen
  - Nationales Centrum für Tumorerkrankungen (NCT), Heidelberg
- St Vincent's University Hospital, Dublin, Ireland
- Italy (5):
  - IRCCS Azienda Ospedaliera Universitaria, San Martino, Genova
  - Azienda Ospedaliera - Universitaria Careggi, Florence
  - Fondacione IRCCS Istituto Nazionale Dei Tumori, Milan
  - Università degli Studi "Federico II" di Napoli, Napoli
  - Azienda Ospedaliera sant'Andrea, Roma
- Netherlands (3):
  - AVL/NKI Medisch Oncologie, Amsterdam
  - Academic Medical Center, Amsterdam
  - Erasmus MC, Rotterdam
- Poland (3):
  - Samodzielny Publiczny Szpital Kliniczny nr 5, Katowice
  - Katedra i Klinika Endokrynologii, Poznan
  - Centrum Diagnostyczno-Lecznicze "GAMMED", Warsaw
- Spain (4):
  - Hospital Universitario Vall D'hebron, Barcelona
  - Hospital Universitario Ramón Y Cajal, Madrid
  - Hospital Universitario 12 De Octubre, Madrid
  - Hospital Universitario Central de Asturias, Oviedo
- United Kingdom (3):
  - Queen Elizabeth Medical Center, Birmingham
  - Royal Free Hospital, London
  - The Christie Hospital NHS Foundation Trust, Manchester

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects with well differentiated, metastatic or locally advanced, unresectable, pancreatic or midgut neuroendocrine tumours (NETs) and who had radiologically documented disease progression as per Response Evaluation Criteria in Solid Tumours (RECIST) v1.0 whilst receiving treatment with lanreotide Autogel® 120mg, every 28 days for at least 24 weeks were enrolled into this study in 25 centres across 10 countries.
Pre-assignment Details: Subjects who had centrally reviewed, radiologically documented disease progression within 24 months prior to enrolment and whilst receiving treatment with lanreotide Autogel® 120 mg, administered every 28 days for at least 24 weeks, were recruited into one of two cohorts based on the primary location of NET (i.e. pancreatic NET [panNET] or midgut NET cohort).
Groups:
- Pancreatic NET (panNET) Cohort: Subjects were treated with lanreotide Autogel® 120 mg, administered as deep subcutaneous (SC) injections, every 14 days starting from Day 1 (at a reduced dosing interval) for up to 48 weeks or until disease progression, death or unacceptable toxicity or tolerability. Subjects who had not progressed at Week 48 could continue study treatment with lanreotide Autogel® 120 mg every 14 days until 25 events (progressive disease [PD] or death) in the panNET cohort had been observed. Additional visits were performed every 12 weeks until disease progression or death, or unacceptable toxicity or tolerability.
- Midgut NET Cohort: Subjects were treated with lanreotide Autogel® 120 mg, administered as deep SC injections, every 14 days starting from Day 1 (at a reduced dosing interval) for up to 96 weeks or until disease progression, death or unacceptable toxicity or tolerability. Subjects who had not progressed at Week 96 could continue study treatment with lanreotide Autogel® 120 mg every 14 days until 25 events (PD or death) in the midgut NET cohort had been observed. Additional visits were performed every 12 weeks until disease progression or death, or unacceptable toxicity or tolerability.
Period: Overall Study
Arm/Group | Pancreatic NET (panNET) Cohort | Midgut NET Cohort
Started | 48 | 51
Completed | 43 | 46
Not Completed | 5 | 5
Not completed — Adverse Event | 2 | 2
Not completed — Consent Withdrawn | 2 | 0
Not completed — Local PD | 0 | 2
Not completed — Investigator Decision | 1 | 1

BASELINE CHARACTERISTICS:
Population: The full analysis set (FAS) included all subjects who received at least one dose of lanreotide Autogel® 120 mg every 14 days during the study.
Groups:
- PanNET Cohort: Subjects were treated with lanreotide Autogel® 120 mg, administered as deep SC injections, every 14 days starting from Day 1 (at a reduced dosing interval) for up to 48 weeks or until disease progression, death or unacceptable toxicity or tolerability. Subjects who had not progressed at Week 48 could continue study treatment with lanreotide Autogel® 120 mg every 14 days until 25 events (PD or death) in the panNET cohort had been observed. Additional visits were performed every 12 weeks until disease progression or death, or unacceptable toxicity or tolerability.
- Total: Total of all reporting groups
Arm/Group | PanNET Cohort | Midgut NET Cohort | Total
Number analyzed (Participants) | 48 | 51 | 99
Age, Continuous [Mean (Standard Deviation); unit: years] | 63.3 (10.6) | 67.1 (8.2) | 65.2 (9.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 28 | 22 | 50
  Male | 20 | 29 | 49
Race/Ethnicity, Customized [Count of Participants; unit: Participants] — Population: French local regulation does not allow the collection of race and therefore French subjects are not included in this baseline measure.
  Participants
    Race: number analyzed (Participants) | 36 | 38 | 74
    Race: Asian | 0 | 1 | 1
    Race: White | 35 | 37 | 72
    Race: Other | 1 | 0 | 1
Region of Enrollment [Number; unit: participants]
  Netherlands | 1 | 3 | 4
  Belgium | 3 | 2 | 5
  Ireland | 2 | 0 | 2
  Denmark | 1 | 2 | 3
  Poland | 12 | 10 | 22
  Italy | 2 | 6 | 8
  United Kingdom | 6 | 9 | 15
  France | 12 | 13 | 25
  Germany | 8 | 3 | 11
  Spain | 1 | 3 | 4
Quality of Life (QoL) Questionnaire Core 30 (QLQ-C30) Score [Mean (Standard Deviation); unit: score on a scale] — QoL was measured Using European Organisation Into the Research and Treatment of Cancer (EORTC), QLQ-C30 v3.0. The global health status sub-score was assessed using the last 2 questions which represented subject's assessment of overall health & QoL. Each question was coded on a 7-point scale (1=very poor to 7=excellent). The sub-score was transformed to range from 0-100, with a high score for global health status representing a high QoL. Population: Only subjects who had a QLQ-C30 measure at baseline are included.
  score on a scale
    number analyzed (Participants) | 46 | 50 | 96
    (all) | 68.12 (19.74) | 67.83 (20.76) | 67.97 (20.17)
EuroQoL 5 Dimensions, 5 Levels (EQ-5D-5L) v1.0 Questionnaire Descriptive System Score [Mean (Standard Deviation); unit: score on a scale] — The EQ-5D-5L descriptive system comprised the following 5 dimensions: mobility, self-care, usual activities, pain/discomfort and anxiety/depression. Each dimension had 5 levels: no problems, slight problems, moderate problems, severe problems, extreme problems. The EQ-5D-5L health states, defined by the EQ-5D-5L descriptive system, was converted into a single index value with scores ranging from 0 (no problems) to 1 (extreme problems). Population: Only subjects with a EQ-5D-5L index value at baseline are included.
  score on a scale
    number analyzed (Participants) | 45 | 45 | 90
    (all) | 0.82 (0.17) | 0.83 (0.14) | 0.83 (0.15)
EQ-5D-5L Visual Analogue Scale (VAS) Score [Mean (Standard Deviation); unit: score on a scale] — The EQ-5D-5L VAS recorded the subject's self-rated health on a vertical VAS which is numbered from 0 (worst health state) to 100 (best health state). Population: Only subjects with a EQ-5D-5L VAS score at baseline are included.
  score on a scale
    number analyzed (Participants) | 47 | 44 | 91
    (all) | 75.02 (17.93) | 70.45 (14.93) | 72.81 (16.62)
QoL Questionnaire Gastrointestinal Neuroendocrine Tumour 21 (QLQ-GI.NET21) Score [Mean (Standard Deviation); unit: score on a scale] — The EORTC QLQ-GI.NET21 module comprised 21 questions that used a 4-point scale (1 = Not at all, 2 = A little, 3 = Quite a bit, 4 = Very much) to evaluate 3 defined multi-item symptom scales (endocrine, gastrointestinal and treatment related side effects), 2 single item symptoms (bone/muscle pain and concern about weight loss), 2 psychosocial scales (social function and disease-related worries) and 2 single items (sexuality and communication). Answers were converted on a grading scale and then individual sub-scores transformed to range from 0 to 100 with a higher score = more or worse problems. Population: Only subjects who had a QLQ GI.NET21 measure at baseline are included.
  score on a scale
    Endocrine Symptoms: number analyzed (Participants) | 45 | 49 | 94
    Endocrine Symptoms | 16.54 (22.30) | 19.73 (22.82) | 18.20 (22.51)
    Gastrointestinal Symptoms: number analyzed (Participants) | 45 | 49 | 94
    Gastrointestinal Symptoms | 21.70 (20.01) | 22.04 (17.17) | 21.88 (18.48)
    Treatment Related Symptoms: number analyzed (Participants) | 32 | 32 | 64
    Treatment Related Symptoms | 11.63 (13.11) | 11.46 (13.75) | 11.55 (13.33)
    Social Function: number analyzed (Participants) | 45 | 49 | 94
    Social Function | 32.84 (24.18) | 35.03 (24.33) | 33.98 (24.15)
    Disease Related Worries: number analyzed (Participants) | 45 | 49 | 94
    Disease Related Worries | 44.44 (29.96) | 44.22 (25.83) | 44.33 (27.74)
    Muscle/Bone Pain: number analyzed (Participants) | 44 | 48 | 92
    Muscle/Bone Pain | 26.52 (30.99) | 25.69 (30.16) | 26.09 (30.39)
    Sexual Function: number analyzed (Participants) | 31 | 28 | 59
    Sexual Function | 22.58 (30.29) | 17.86 (27.94) | 20.34 (29.04)
    Information/Communication Function: number analyzed (Participants) | 45 | 48 | 93
    Information/Communication Function | 3.70 (12.76) | 4.17 (11.14) | 3.94 (11.89)
    Body Image: number analyzed (Participants) | 44 | 45 | 89
    Body Image | 10.61 (23.60) | 15.56 (28.95) | 13.11 (26.41)
Categories of Proliferation index Ki67 [Number; unit: participants]
  ≥10% | 7 | 4 | 11
  <10% | 41 | 46 | 87
  Missing | 0 | 1 | 1
Tumour grading (according to WHO 2010 classification) [Number; unit: participants] — According to the 2010 WHO classification, Grade 1 NET is defined as <=2% Ki-67 labelling index; and Grade 2 NET is defined as 3-20% Ki-67 labelling index. Grade 2 is considered to have a worse outcome.
  participants
    Grade 1 | 12 | 29 | 41
    Grade 2 | 36 | 22 | 58
Hepatic tumour load [Number; unit: participants]
  >25% | 7 | 9 | 16
  ≤25% | 41 | 42 | 83

OUTCOME MEASURES:

1. Primary Outcome: Median Progression Free Survival (PFS)
Description: PFS was defined as the time from first injection of lanreotide Autogel® 120 mg every 14 days to progression or death. Disease progression was assessed by tumour response evaluation according to RECIST v1.0, every 12 weeks, measured by independent central review using the same imaging technique (computed tomography [CT] scan or magnetic resonance imaging [MRI]) for each subject throughout the study. The median PFS time was estimated using the Kaplan Meier method for each cohort.
Time Frame: From Day 1 up to Week 60 for the panNET cohort and Week 103 for the midgut NET cohort
Population: The FAS included all subjects who received at least one dose of lanreotide Autogel® 120 mg every 14 days during the study.
Measure: Median (95% Confidence Interval); unit: months
Groups:
- PanNET Cohort: Subjects were treated with lanreotide Autogel® 120 mg, administered as SC injections, every 14 days starting from Day 1 (at a reduced dosing interval) for up to 48 weeks or until disease progression, death or unacceptable toxicity or tolerability. Subjects who had not progressed at Week 48 could continue study treatment with lanreotide Autogel® 120 mg every 14 days until 25 events (PD or death) in the panNET cohort had been observed. Additional visits were performed every 12 weeks until disease progression or death, or unacceptable toxicity or tolerability.
Arm/Group | PanNET Cohort | Midgut NET Cohort
Number analyzed (Participants) | 48 | 51
months | 5.6 [5.5 to 8.3] | 8.3 [5.6 to 11.1]

2. Secondary Outcome: Median Time to Progression
Description: Time to Progression was defined as time from first injection of lanreotide Autogel® 120 mg every 14 days to progression. Disease progression was assessed by tumour response evaluation according to RECIST v1.0, every 12 weeks, measured by independent central review using the same imaging technique (CT scan or MRI) for each subject throughout the study. Median time to progression was estimated using the Kaplan Meier method for each cohort.
Time Frame: From Day 1 up to Week 60 for the panNET cohort and Week 103 for the midgut NET cohort
Population: as for outcome 1
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | PanNET Cohort | Midgut NET Cohort
Number analyzed (Participants) | 48 | 51
months | 5.6 [5.5 to 8.3] | 8.7 [8.3 to 13.9]

3. Secondary Outcome: Percentage of Subjects Alive and Progression Free
Description: The percentage of subjects alive and progression-free was assessed throughout the study up to Week 60 for the panNET cohort and Week 96 for the midgut cohort. Disease progression was assessed by tumour response evaluation according to RECIST v1.0, every 12 weeks measured by independent central review using the same imaging technique (CT scan or MRI) for each subject throughout the study. The percentage of subjects alive and progression free was estimated using the Kaplan Meier method for each cohort.
Time Frame: Weeks 12, 24, 36, 48, 60 (for both cohorts) and Weeks 72, 84 and 96 (for midgut NET cohort)
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: percentage of subjects
Arm/Group | PanNET Cohort | Midgut NET Cohort
Number analyzed (Participants) | 48 | 51
percentage of subjects
  Week 12 | 93.3 [80.7 to 97.8] | 91.8 [79.7 to 96.9]
  Week 24 | 64.4 [48.7 to 76.5] | 65.3 [50.3 to 76.8]
  Week 36 | 37.8 [23.9 to 51.6] | 59.2 [44.2 to 71.4]
  Week 48 | 28.5 [16.2 to 42.1] | 38.3 [24.8 to 51.6]
  Week 60 | 20.7 [9.0 to 35.7] | 36.1 [22.9 to 49.5]
  Week 72: number analyzed (Participants) | 0 | 51
  Week 72 |  | 29.8 [17.6 to 42.9]
  Week 84: number analyzed (Participants) | 0 | 51
  Week 84 |  | 27.5 [15.7 to 40.5]
  Week 96: number analyzed (Participants) | 0 | 51
  Week 96 |  | 25.2 [13.9 to 38.1]

4. Secondary Outcome: Overall Survival
Description: Overall survival was defined as the time in months from the first injection of lanreotide Autogel® 120 mg every 14 days to death due to any cause. Median overall survival was estimated using the Kaplan Meier method for each cohort.
Time Frame: From Day 1 up to Week 60 for the panNET cohort and Week 103 for the midgut NET cohort
Population: as for outcome 1
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | PanNET Cohort | Midgut NET Cohort
Number analyzed (Participants) | 48 | 51
months | NA [NA to NA] — The median overall survival from the Kaplan Meier model was not reached for this cohort. | NA [NA to NA] — The median overall survival from the Kaplan Meier model was not reached for this cohort.

5. Secondary Outcome: Objective Response Rate (ORR)
Description: The ORR was defined as the percentage of subjects who achieve either complete response (CR) or partial response (PR) according to RECIST v1.0 criteria. ORR was evaluated every 12 weeks and results are presented for each cohort.
Time Frame: Weeks 12, 24, 36, 48, 60 (for both cohorts) and Weeks 72, 84, and 96 (for midgut cohort)
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: percentage of subjects
Arm/Group | PanNET Cohort | Midgut NET Cohort
Number analyzed (Participants) | 48 | 51
percentage of subjects
  Week 12 | 0.0 [0.0 to 7.4] | 0.0 [0.0 to 7.0]
  Week 24 | 0.0 [0.0 to 7.4] | 0.0 [0.0 to 7.0]
  Week 36 | 0.0 [0.0 to 7.4] | 0.0 [0.0 to 7.0]
  Week 48 | 0.0 [0.0 to 7.4] | 0.0 [0.0 to 7.0]
  Week 60 | 0.0 [0.0 to 7.4] | 2.0 [0.0 to 10.4]
  Week 72: number analyzed (Participants) | 0 | 51
  Week 72 |  | 3.9 [0.5 to 13.5]
  Week 84: number analyzed (Participants) | 0 | 51
  Week 84 |  | 2.0 [0.0 to 10.4]
  Week 96: number analyzed (Participants) | 0 | 51
  Week 96 |  | 2.0 [0.0 to 10.4]

6. Secondary Outcome: Disease Control Rate (DCR)
Description: The DCR was defined as the percentage of subjects who achieved CR plus PR plus Stable Disease (SD), evaluated according to RECIST v1.0 criteria. The DCR at Weeks 24 and 48 is presented for each cohort.
Time Frame: Weeks 24 and 48
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: percentage of subjects
Arm/Group | PanNET Cohort | Midgut NET Cohort
Number analyzed (Participants) | 48 | 51
percentage of subjects
  Week 24 | 43.8 [29.5 to 58.8] | 58.8 [44.2 to 72.4]
  Week 48 | 22.9 [12.0 to 37.3] | 33.3 [20.8 to 47.9]

7. Secondary Outcome: Best Overall Response Rate
Description: Best overall response was defined as the best response recorded from the initiation of treatment until disease progression, according to RECIST v1.0 evaluation. The percentage of subjects in each response category and those who were non-evaluable (i.e. with no tumour assessment after the start of study treatment) throughout the study are presented for each cohort.
Time Frame: From Day 1 up to Week 60 for the panNET cohort and Week 103 for the midgut NET cohort
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: percentage of subjects
Arm/Group | PanNET Cohort | Midgut NET Cohort
Number analyzed (Participants) | 48 | 51
percentage of subjects
  CR | 0.0 [0.0 to 7.4] | 0.0 [0.0 to 7.0]
  PR | 0.0 [0.0 to 7.4] | 3.9 [0.5 to 13.5]
  SD | 66.7 [51.6 to 79.6] | 68.6 [54.1 to 80.9]
  PD | 31.3 [18.7 to 46.3] | 23.5 [12.8 to 37.5]
  Not evaluable | 0.0 [0.0 to 7.4] | 2.0 [0.0 to 10.4]

8. Secondary Outcome: Median Duration of Stable Disease
Description: Median duration of SD was the time from first injection of lanreotide Autogel® 120 mg every 14 days until the first occurrence of PD by central assessment. Disease progression was assessed by tumour response evaluation according to RECIST v1.0, every 12 weeks, measured using the same imaging technique (CT scan or MRI) for each subject throughout the study. Median duration of stable disease was estimated using the Kaplan Meier method for each cohort.
Time Frame: From Day 1 up to Week 60 for the panNET cohort and Week 103 for the midgut NET cohort
Population: as for outcome 1
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | PanNET Cohort | Midgut NET Cohort
Number analyzed (Participants) | 48 | 51
months | 8.3 [8.0 to 13.8] | 13.8 [8.6 to NA] — 95% confidence interval upper limit could not be calculated as an insufficient number of events were observed.

9. Secondary Outcome: Factors Associated With PFS
Description: A univariate cox proportional hazards model was used to assess whether the following factors were associated with PFS:
  * Hepatic tumour load: >25% versus reference ≤25%
  * Tumour Grade: Grade 2 versus reference Grade 1,
  * Previous surgery of the primary tumour: No versus reference Yes,
  * Proliferation index Ki67: ≥10% versus reference <10%
  * Duration of treatment with lanreotide Autogel® 120 mg every 28 days by category: ≥median value versus reference <median value,
  * Age by category: ≥65 years versus reference <65 years,
  * Time from diagnosis to study entry by category: ≥3 years versus reference <3 years,
  * Time interval between the two CT scans (pre-screening/screening): ≥12 months versus reference <12 months and
  * Symptoms (diarrhoea or flushing at baseline): No versus reference Yes.
  Each factor was assessed for its importance in the Cox model for PFS in a univariate fashion.
Time Frame: Screening/Baseline (Day 1)
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Hazard Ratio
Arm/Group | PanNET Cohort | Midgut NET Cohort
Number analyzed (Participants) | 48 | 51
Hazard Ratio
  Hepatic tumour load: >25% Vs ≤25% | 0.96 [0.40 to 2.32] | 1.54 [0.70 to 3.40]
  Tumour Grade: 2 Vs 1 | 0.68 [0.32 to 1.45] | 0.90 [0.46 to 1.77]
  Previous surgery: No Vs Yes | 1.04 [0.53 to 2.04] | 2.14 [0.83 to 5.52]
  Ki67: ≥10% Vs <10%: number analyzed (Participants) | 48 | 50
  Ki67: ≥10% Vs <10% | 3.60 [1.39 to 9.32] | 2.26 [0.67 to 7.60]
  Duration of treatment with lanreotide Autogel® 120 mg every 28 days: ≥median Vs <median | 0.68 [0.34 to 1.34] | 0.76 [0.40 to 1.47]
  Age: ≥65 years Vs <65 years | 1.55 [0.79 to 3.06] | 1.15 [0.58 to 2.31]
  Time from diagnosis: ≥3 years Vs <3 years | 0.49 [0.25 to 0.96] | 0.94 [0.49 to 1.82]
  Time between CT scans: ≥12 months Vs <12 months | 0.47 [0.24 to 0.94] | 0.72 [0.37 to 1.39]
  Symptoms: No Vs Yes: number analyzed (Participants) | 48 | 50
  Symptoms: No Vs Yes | 2.55 [0.89 to 7.28] | 1.32 [0.68 to 2.56]

10. Secondary Outcome: Mean Change From Baseline in Number of Stools and Flushing Episodes
Description: Symptom control was measured by the total number of stools (diarrhoea) and flushing episodes during the 7 days prior to the visit, reported orally by the subject to the investigator. The mean change from baseline in number of stools and flushing episodes reported at each visit is presented for each cohort.
Time Frame: Baseline (Day 1), Weeks 8,12, 48 and end of study (approximately 64 weeks for panNET cohort and 108 weeks for midgut NET cohort)
Population: The FAS included all subjects who received at least one dose of lanreotide Autogel® 120 mg every 14 days during the study. Numbers analysed at each time point correspond to the number of subjects reporting episodes in the 7 days prior to the visit.
Measure: Mean (Standard Deviation); unit: episodes
Arm/Group | PanNET Cohort | Midgut NET Cohort
Number analyzed (Participants) | 48 | 51
episodes
  Stools - Week 8: number analyzed (Participants) | 5 | 13
  Stools - Week 8 | 1.0 (5.5) | -1.0 (8.2)
  Stools - Week 12: number analyzed (Participants) | 5 | 13
  Stools - Week 12 | -1.2 (7.9) | 0.7 (2.5)
  Stools - Week 48: number analyzed (Participants) | 2 | 5
  Stools - Week 48 | -1.0 (0.0) | 3.4 (4.8)
  Stools - End of Study: number analyzed (Participants) | 4 | 5
  Stools - End of Study | 0.5 (5.4) | -1.2 (12.2)
  Flushing - Week 8: number analyzed (Participants) | 3 | 9
  Flushing - Week 8 | 0.7 (2.1) | -3.3 (8.3)
  Flushing - Week 12: number analyzed (Participants) | 2 | 6
  Flushing - Week 12 | -1.0 (0.0) | 1.5 (10.0)
  Flushing - Week 48: number analyzed (Participants) | 2 | 2
  Flushing - Week 48 | -1.0 (0.0) | -1.5 (2.1)
  Flushing - End of Study: number analyzed (Participants) | 2 | 4
  Flushing - End of Study | 0.0 (1.4) | -0.5 (6.2)

11. Secondary Outcome: Mean Change From Baseline in QoL Measured Using EORTC, QLQ-C30 v3.0 (Global Health Status Sub-score)
Description: Subjects were instructed to complete the 30 questions in the EORTC-QLQ-C30 v3.0 questionnaire at baseline and every 12 weeks throughout the study.
  The global health status sub-score was assessed using the last 2 questions which represented subject's assessment of overall health & QoL. Each question was coded on a 7-point scale (1=very poor to 7=excellent). The sub-score was transformed to range from 0-100, with a high score for global health status representing a high QoL. The mean change from baseline in the transformed global health status are presented for the end of study/early withdrawal visit, with a positive change indicating an improvement in QoL.
Time Frame: Baseline (Day 1) and end of study (approximately 64 weeks for panNET cohort and 108 weeks for midgut NET (and overall) cohort)
Population: The FAS included all subjects who received at least one dose of lanreotide Autogel® 120 mg every 14 days during the study. Only subjects with data available for analysis are presented.
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- Overall: All subjects who received at least one dose of lanreotide Autogel® 120 mg every 14 days during the study.
Arm/Group | PanNET Cohort | Midgut NET Cohort | Overall
Number analyzed (Participants) | 22 | 25 | 47
score on a scale | -0.38 (15.32) | -1.33 (17.13) | -0.89 (16.14)

12. Secondary Outcome: Mean Change From Baseline in EQ-5D-5L v1.0 Questionnaire (Descriptive System)
Description: Subjects were instructed to complete the EQ-5D-5L descriptive system at baseline and every 12 weeks throughout the study.
  The EQ-5D-5L descriptive system comprised the following 5 dimensions: mobility, self-care, usual activities, pain/discomfort and anxiety/depression. Each dimension had 5 levels: no problems, slight problems, moderate problems, severe problems, extreme problems. The EQ-5D-5L health states, defined by the EQ-5D-5L descriptive system, was converted into a single index value with scores ranging from 0 (no problems) to 1 (extreme problems). The mean change from baseline at the end of study/early withdrawal visit is presented with a positive change from baseline in the index values indicating a worsening of symptoms.
Time Frame: as for outcome 11
Population: as for outcome 11
Measure: Mean (Standard Deviation); unit: Index value
Arm/Group | PanNET Cohort | Midgut NET Cohort | Overall
Number analyzed (Participants) | 22 | 21 | 43
Index value | -0.04 (0.12) | 0.00 (0.11) | -0.02 (0.12)

13. Secondary Outcome: Mean Change From Baseline in EQ-5D-5L v1.0 Questionnaire (VAS)
Description: Subjects were instructed to complete the EQ-5D-5L VAS at baseline and every 12 weeks throughout the study. The EQ-5D-5L VAS recorded the subject's self-rated health on a vertical VAS which is numbered from 0 (worst health state) to 100 (best health state). The mean change from baseline at the end of study/early withdrawal visit is presented with a positive change in the VAS indicating an improvement in symptoms.
Time Frame: as for outcome 11
Population: as for outcome 11
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | PanNET Cohort | Midgut NET Cohort | Overall
Number analyzed (Participants) | 21 | 21 | 42
score on a scale | -1.90 (14.80) | -1.76 (9.34) | -1.83 (12.22)

14. Secondary Outcome: Mean Change From Baseline in QoL Questionnaire Gastrointestinal Neuroendocrine Tumour 21 (QLQ-GI.NET21; 2006)
Description: Subjects were asked to complete the EORTC QLQ-GI.NET21 module which comprised 21 questions that used a 4-point scale (1 = Not at all, 2 = A little, 3 = Quite a bit, 4 = Very much) to evaluate 3 defined multi-item symptom scales (endocrine, gastrointestinal and treatment related side effects), 2 single item symptoms (bone/muscle pain and concern about weight loss), 2 psychosocial scales (social function and disease-related worries) and 2 other single items (sexuality and communication). Answers were converted into grading scale, with values between 0 and 100. Each individual sub-score was transformed to range from 0 to 100. The mean change from baseline at the end of study/early withdrawal visit is presented with a higher score representing more or worse problems.
Time Frame: as for outcome 11
Population: as for outcome 11
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | PanNET Cohort | Midgut NET Cohort | Overall
Number analyzed (Participants) | 48 | 51 | 99
score on a scale
  Endocrine Symptoms: number analyzed (Participants) | 21 | 24 | 45
  Endocrine Symptoms | -0.53 (11.37) | -5.09 (17.33) | -2.96 (14.87)
  Gastrointestinal Symptoms: number analyzed (Participants) | 21 | 24 | 45
  Gastrointestinal Symptoms | -3.49 (14.24) | -2.78 (15.96) | -3.11 (15.02)
  Treatment Related Symptoms: number analyzed (Participants) | 15 | 16 | 31
  Treatment Related Symptoms | 5.93 (15.64) | -3.47 (14.47) | 1.08 (15.54)
  Social Function: number analyzed (Participants) | 21 | 24 | 45
  Social Function | -0.79 (13.41) | -9.49 (18.20) | -5.43 (16.56)
  Disease Related Worries: number analyzed (Participants) | 21 | 24 | 45
  Disease Related Worries | 3.17 (15.47) | -0.93 (27.40) | 0.99 (22.48)
  Muscle/Bone Pain: number analyzed (Participants) | 20 | 24 | 44
  Muscle/Bone Pain | -1.67 (33.29) | 0.00 (36.78) | -0.76 (34.84)
  Sexual Function: number analyzed (Participants) | 14 | 12 | 26
  Sexual Function | 2.38 (15.82) | -2.78 (26.43) | 0.00 (21.08)
  Information/Communication Function: number analyzed (Participants) | 21 | 23 | 44
  Information/Communication Function | 7.94 (29.64) | -2.90 (9.60) | 2.27 (22.04)
  Body Image: number analyzed (Participants) | 20 | 22 | 42
  Body Image | 0.00 (15.29) | -7.58 (28.97) | -3.97 (23.52)

15. Secondary Outcome: Mean Change From Baseline in Nonspecific Tumour Biomarkers
Description: Nonspecific tumour peptide biomarkers (chromogranin A [CgA], neuron specific enolase [NSE] and plasma/urinary 5-hydroxyindoleacetic acid [5-HIAA]) were evaluated in both pancreas and midgut subjects at baseline and Week 12 and every 12 weeks thereafter. At all scheduled visits, except baseline, plasma/urinary 5-HIAA was only performed in subjects with symptoms of carcinoid syndrome (diarrhoea and/or flushing) or if urinary 5-HIAA was elevated (above upper limit of normal [ULN]) at baseline. Mean change from baseline values were normalised by the ULN (xULN) and are presented for each cohort.
Time Frame: Baseline (Day 1) and end of study (approximately 64 weeks for panNET cohort and 108 weeks for midgut NET cohort)
Population: as for outcome 11
Measure: Mean (Standard Deviation); unit: xULN
Arm/Group | PanNET Cohort | Midgut NET Cohort
Number analyzed (Participants) | 48 | 51
xULN
  CgA: number analyzed (Participants) | 22 | 24
  CgA | 0.205 (1.258) | 0.370 (1.843)
  NSE: number analyzed (Participants) | 15 | 10
  NSE | 0.03 (1.00) | -0.49 (1.86)
  Plasma 5-HIAA: number analyzed (Participants) | 20 | 17
  Plasma 5-HIAA | -0.42 (1.44) | 3.90 (7.39)

16. Secondary Outcome: Mean Change From Baseline in PanNet Specific Tumour Biomarkers: Pancreatic Polypeptide, Gastrin
Description: PanNET specific tumour peptide biomarkers were evaluated in pancreas subjects at baseline. Only the tumour biomarkers that were above normal range at baseline were evaluated every 12 weeks thereafter and at the end of study visit. The mean change from baseline values in picomole/liter (pmol/L) are presented for the end of study visit.
Time Frame: Baseline (Day 1) and end of study (approximately 64 weeks)
Population: The FAS included all subjects who received at least one dose of lanreotide Autogel® 120 mg every 14 days during the study. Only subjects in the panNET cohort with data available for analysis are presented.
Measure: Mean (Standard Deviation); unit: pmol/L
Arm/Group | PanNET Cohort
Number analyzed (Participants) | 48
pmol/L
  Pancreatic Polypeptide: number analyzed (Participants) | 3
  Pancreatic Polypeptide | 82.7 (146.7)
  Gastrin: number analyzed (Participants) | 4
  Gastrin | -9.8 (70.7)

17. Secondary Outcome: Mean Change From Baseline in PanNet Specific Tumour Biomarkers: Glucagon
Description: PanNET specific tumour peptide biomarkers were evaluated in pancreas subjects at baseline. Only the tumour biomarkers that were above normal range at baseline were evaluated every 12 weeks thereafter and at the end of study visit. The mean change from baseline values in nanograms (ng)/L are presented for the end of study visit.
Time Frame: Baseline (Day 1) and end of study (approximately 64 weeks)
Population: The FAS included all subjects who received at least one dose of lanreotide Autogel® 120 mg every 14 days during the study. Only subjects in panNET cohort with data available for analysis are presented.
Measure: Mean (Standard Deviation); unit: ng/L
Arm/Group | PanNET Cohort
Number analyzed (Participants) | 4
ng/L | 5.5 (36.4)

ADVERSE EVENTS:
Time Frame: Treatment emergent adverse events were recorded from the first dose of lanreotide Autogel® 120 mg on Day 1 until 28 days after the last treatment. Overall time frame of up to a maximum of 64 weeks for panNET cohort and 108 weeks for midgut NET (and overall) cohort.
Description: The FAS included all subjects who received at least one dose of lanreotide Autogel® 120 mg every 14 days during the study.
Groups:
- Overall Subjects: All subjects who received at least one dose of lanreotide Autogel® 120 mg every 14 days during the study.
Arm/Group | PanNET Cohort | Midgut NET Cohort | Overall Subjects
All-Cause Mortality (participants affected / at risk) | 1/48 | 3/51 | 4/99
Serious Adverse Events (participants affected / at risk) | 5/48 | 13/51 | 18/99
Other Adverse Events (participants affected / at risk) | 41/48 | 47/51 | 88/99
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | PanNET Cohort (N=48) | Midgut NET Cohort (N=51) | Overall Subjects (N=99)
Cardiac failure (Cardiac disorders) | 0 (0) | 1 (1) | 1 (1)
Pulseless electrical activity (Cardiac disorders) | 0 (0) | 1 (1) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 1 (2) | 1 (2)
Diarrhoea (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1)
Intestinal obstruction (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1)
Asthenia (General disorders) | 0 (0) | 1 (1) | 1 (1)
Chest pain (General disorders) | 0 (0) | 1 (1) | 1 (1)
General physical health deterioration (General disorders) | 0 (0) | 1 (1) | 1 (1)
Anaphylactic reaction (Immune system disorders) | 1 (1) | 0 (0) | 1 (1)
Peritonitis (Infections and infestations) | 0 (0) | 1 (1) | 1 (1)
Viral infection (Infections and infestations) | 0 (0) | 1 (1) | 1 (1)
Craniocerebral injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 1 (1)
Fall (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 1 (1)
Spinal fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 1 (1)
Bone neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 1 (1)
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 1 (1)
Spinal cord compression (Nervous system disorders) | 0 (0) | 1 (1) | 1 (1)
Syncope (Nervous system disorders) | 1 (1) | 0 (0) | 1 (1)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (3) | 3 (4)
Hypotension (Vascular disorders) | 0 (0) | 1 (1) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | PanNET Cohort (N=48) | Midgut NET Cohort (N=51) | Overall Subjects (N=99)
Lymphopenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 1 (1)
Monocytopenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 1 (1)
Arrhythmia (Cardiac disorders) | 1 (1) | 0 (0) | 1 (1)
Cardiac failure (Cardiac disorders) | 0 (0) | 1 (2) | 1 (2)
Heart valve incompetence (Cardiac disorders) | 0 (0) | 1 (1) | 1 (1)
Palpitations (Cardiac disorders) | 1 (1) | 0 (0) | 1 (1)
Right ventricular failure (Cardiac disorders) | 0 (0) | 1 (1) | 1 (1)
Tachycardia (Cardiac disorders) | 1 (1) | 0 (0) | 1 (1)
Tricuspid valve disease (Cardiac disorders) | 0 (0) | 1 (1) | 1 (1)
Deafness (Ear and labyrinth disorders) | 1 (1) | 0 (0) | 1 (1)
Deafness unilateral (Ear and labyrinth disorders) | 1 (1) | 0 (0) | 1 (1)
Ear pain (Ear and labyrinth disorders) | 0 (0) | 1 (1) | 1 (1)
Hypoacusis (Ear and labyrinth disorders) | 1 (1) | 0 (0) | 1 (1)
Vertigo (Ear and labyrinth disorders) | 0 (0) | 1 (2) | 1 (2)
Vertigo positional (Ear and labyrinth disorders) | 1 (1) | 0 (0) | 1 (1)
Diplopia (Eye disorders) | 0 (0) | 1 (1) | 1 (1)
Dry eye (Eye disorders) | 0 (0) | 1 (1) | 1 (1)
Eye pain (Eye disorders) | 0 (0) | 1 (1) | 1 (1)
Eye pruritus (Eye disorders) | 0 (0) | 1 (1) | 1 (1)
Glaucoma (Eye disorders) | 0 (0) | 1 (1) | 1 (1)
Ocular hyperaemia (Eye disorders) | 0 (0) | 2 (2) | 2 (2)
Abdominal discomfort (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1)
Abdominal distension (Gastrointestinal disorders) | 0 (0) | 6 (7) | 6 (7)
Abdominal pain (Gastrointestinal disorders) | 7 (13) | 12 (16) | 19 (29)
Abdominal pain lower (Gastrointestinal disorders) | 1 (1) | 1 (1) | 2 (2)
Abdominal pain upper (Gastrointestinal disorders) | 2 (2) | 6 (7) | 8 (9)
Anal incontinence (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1)
Anorectal discomfort (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1)
Ascites (Gastrointestinal disorders) | 0 (0) | 2 (2) | 2 (2)
Constipation (Gastrointestinal disorders) | 2 (3) | 2 (3) | 4 (6)
Diarrhoea (Gastrointestinal disorders) | 14 (20) | 27 (35) | 41 (55)
Dry mouth (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1)
Dyspepsia (Gastrointestinal disorders) | 0 (0) | 2 (3) | 2 (3)
Faeces discoloured (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1)
Flatulence (Gastrointestinal disorders) | 1 (1) | 6 (8) | 7 (9)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1 (1) | 2 (2) | 3 (3)
Gingival bleeding (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1)
Gingival pain (Gastrointestinal disorders) | 1 (1) | 1 (1) | 2 (2)
Glossodynia (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1)
Haematochezia (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1)
Hernial eventration (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1)
Inguinal hernia (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1)
Nausea (Gastrointestinal disorders) | 5 (5) | 6 (9) | 11 (14)
Oral pain (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1)
Pancreatic failure (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1)
Proctalgia (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1)
Steatorrhoea (Gastrointestinal disorders) | 2 (2) | 3 (3) | 5 (5)
Stomatitis (Gastrointestinal disorders) | 1 (1) | 1 (1) | 2 (2)
Toothache (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1)
Vomiting (Gastrointestinal disorders) | 6 (9) | 4 (4) | 10 (13)
Asthenia (General disorders) | 4 (24) | 4 (5) | 8 (29)
Chest pain (General disorders) | 0 (0) | 3 (3) | 3 (3)
Fatigue (General disorders) | 7 (8) | 8 (11) | 15 (19)
Gait disturbance (General disorders) | 0 (0) | 1 (1) | 1 (1)
Hunger (General disorders) | 0 (0) | 1 (1) | 1 (1)
Influenza like illness (General disorders) | 1 (1) | 3 (3) | 4 (4)
Injection site bruising (General disorders) | 1 (1) | 0 (0) | 1 (1)
Injection site pain (General disorders) | 0 (0) | 1 (1) | 1 (1)
Malaise (General disorders) | 1 (1) | 2 (2) | 3 (3)
Medical device site pain (General disorders) | 1 (1) | 0 (0) | 1 (1)
Oedema peripheral (General disorders) | 2 (2) | 2 (2) | 4 (4)
Pain (General disorders) | 0 (0) | 1 (1) | 1 (1)
Peripheral swelling (General disorders) | 0 (0) | 3 (3) | 3 (3)
Polyp (General disorders) | 0 (0) | 1 (1) | 1 (1)
Pyrexia (General disorders) | 2 (2) | 2 (5) | 4 (7)
Bile duct stone (Hepatobiliary disorders) | 0 (0) | 1 (1) | 1 (1)
Cholelithiasis (Hepatobiliary disorders) | 0 (0) | 3 (3) | 3 (3)
Hepatic failure (Hepatobiliary disorders) | 0 (0) | 1 (1) | 1 (1)
Liver injury (Hepatobiliary disorders) | 1 (1) | 0 (0) | 1 (1)
Drug hypersensitivity (Immune system disorders) | 0 (0) | 1 (1) | 1 (1)
Bronchitis (Infections and infestations) | 0 (0) | 1 (1) | 1 (1)
Carbuncle (Infections and infestations) | 0 (0) | 1 (1) | 1 (1)
Cystitis (Infections and infestations) | 2 (2) | 1 (1) | 3 (3)
Cystitis bacterial (Infections and infestations) | 0 (0) | 1 (1) | 1 (1)
Diverticulitis (Infections and infestations) | 0 (0) | 2 (2) | 2 (2)
Folliculitis (Infections and infestations) | 0 (0) | 1 (1) | 1 (1)
Herpes zoster (Infections and infestations) | 0 (0) | 2 (2) | 2 (2)
Influenza (Infections and infestations) | 2 (2) | 3 (6) | 5 (8)
Lower respiratory tract infection (Infections and infestations) | 1 (2) | 3 (3) | 4 (5)
Nasopharyngitis (Infections and infestations) | 7 (7) | 5 (6) | 12 (13)
Respiratory tract infection (Infections and infestations) | 0 (0) | 1 (1) | 1 (1)
Tonsillitis (Infections and infestations) | 1 (1) | 0 (0) | 1 (1)
Upper respiratory tract infection (Infections and infestations) | 0 (0) | 1 (1) | 1 (1)
Urinary tract infection (Infections and infestations) | 4 (6) | 1 (1) | 5 (7)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 1 (1)
Incision site pain (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 1 (1)
Incisional hernia (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 1 (1)
Ligament sprain (Injury, poisoning and procedural complications) | 0 (0) | 2 (2) | 2 (2)
Muscle strain (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 1 (1)
Post procedural complication (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 1 (1)
Radiation skin injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 1 (1)
Skin abrasion (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 1 (1)
Alanine aminotransferase increased (Investigations) | 1 (1) | 2 (2) | 3 (3)
Aspartate aminotransferase abnormal (Investigations) | 1 (1) | 0 (0) | 1 (1)
Aspartate aminotransferase increased (Investigations) | 1 (1) | 1 (1) | 2 (2)
Bacterial test positive (Investigations) | 0 (0) | 1 (1) | 1 (1)
Blood alkaline phosphatase increased (Investigations) | 3 (3) | 1 (1) | 4 (4)
Blood bilirubin increased (Investigations) | 0 (0) | 2 (2) | 2 (2)
Blood chromogranin A increased (Investigations) | 0 (0) | 1 (1) | 1 (1)
Blood creatinine increased (Investigations) | 1 (1) | 0 (0) | 1 (1)
Blood glucose decreased (Investigations) | 0 (0) | 1 (1) | 1 (1)
Blood glucose increased (Investigations) | 1 (1) | 1 (1) | 2 (2)
Blood potassium increased (Investigations) | 1 (1) | 0 (0) | 1 (1)
Blood triglycerides increased (Investigations) | 0 (0) | 1 (1) | 1 (1)
Blood urea increased (Investigations) | 1 (1) | 1 (1) | 2 (2)
Blood urine present (Investigations) | 0 (0) | 1 (1) | 1 (1)
C-reactive protein increased (Investigations) | 0 (0) | 1 (1) | 1 (1)
Gamma-glutamyltransferase abnormal (Investigations) | 1 (1) | 0 (0) | 1 (1)
Gamma-glutamyltransferase decreased (Investigations) | 0 (0) | 1 (1) | 1 (1)
Gamma-glutamyltransferase increased (Investigations) | 1 (1) | 2 (2) | 3 (3)
Glycosylated haemoglobin increased (Investigations) | 1 (1) | 0 (0) | 1 (1)
Lymphocyte count decreased (Investigations) | 0 (0) | 1 (1) | 1 (1)
Neutrophil count decreased (Investigations) | 0 (0) | 1 (1) | 1 (1)
Platelet count decreased (Investigations) | 0 (0) | 1 (1) | 1 (1)
Specific gravity urine increased (Investigations) | 1 (1) | 0 (0) | 1 (1)
Urine ketone body present (Investigations) | 2 (2) | 0 (0) | 2 (2)
Weight decreased (Investigations) | 1 (1) | 2 (2) | 3 (3)
Carbohydrate intolerance (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 1 (1)
Decreased appetite (Metabolism and nutrition disorders) | 5 (5) | 2 (2) | 7 (7)
Hypercholesterolaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 1 (1)
Hyperglycaemia (Metabolism and nutrition disorders) | 1 (1) | 1 (1) | 2 (2)
Hyperkalaemia (Metabolism and nutrition disorders) | 0 (0) | 2 (2) | 2 (2)
Hypernatraemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 1 (1)
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 1 (1)
Hyperuricaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 1 (1)
Hypoalbuminaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 1 (1)
Hypocalcaemia (Metabolism and nutrition disorders) | 1 (1) | 2 (2) | 3 (3)
Hypoglycaemia (Metabolism and nutrition disorders) | 1 (3) | 1 (1) | 2 (4)
Hypokalaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 1 (1)
Hyponatraemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 1 (1)
Malnutrition (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 1 (1)
Vitamin D deficiency (Metabolism and nutrition disorders) | 1 (1) | 1 (1) | 2 (2)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 5 (7) | 5 (7)
Back pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 2 (2) | 4 (4)
Exostosis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 1 (1)
Flank pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 1 (1)
Intervertebral disc degeneration (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 1 (1)
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 1 (1)
Joint swelling (Musculoskeletal and connective tissue disorders) | 0 (0) | 3 (5) | 3 (5)
Mobility decreased (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 1 (1)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1 (1) | 2 (3) | 3 (4)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) | 2 (2)
Musculoskeletal discomfort (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 1 (1)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 2 (2) | 3 (3)
Myalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (2) | 1 (2)
Neck pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2) | 2 (2)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) | 2 (2)
Osteoporosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 1 (1)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 2 (2) | 1 (2) | 3 (4)
Periarthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 1 (1)
Rheumatoid arthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (2) | 1 (2)
Spinal pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 2 (2) | 3 (3)
Metastases to liver (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 1 (1)
Ageusia (Nervous system disorders) | 1 (1) | 0 (0) | 1 (1)
Aphasia (Nervous system disorders) | 0 (0) | 1 (2) | 1 (2)
Balance disorder (Nervous system disorders) | 0 (0) | 1 (1) | 1 (1)
Dizziness (Nervous system disorders) | 3 (3) | 5 (7) | 8 (10)
Dizziness postural (Nervous system disorders) | 0 (0) | 1 (1) | 1 (1)
Head discomfort (Nervous system disorders) | 0 (0) | 1 (1) | 1 (1)
Headache (Nervous system disorders) | 3 (3) | 4 (5) | 7 (8)
Lethargy (Nervous system disorders) | 1 (1) | 1 (1) | 2 (2)
Poor quality sleep (Nervous system disorders) | 1 (1) | 1 (1) | 2 (2)
Presyncope (Nervous system disorders) | 0 (0) | 2 (2) | 2 (2)
Sciatica (Nervous system disorders) | 0 (0) | 2 (2) | 2 (2)
Syncope (Nervous system disorders) | 1 (1) | 0 (0) | 1 (1)
Taste disorder (Nervous system disorders) | 1 (1) | 0 (0) | 1 (1)
Tremor (Nervous system disorders) | 1 (1) | 2 (2) | 3 (3)
Acrophobia (Psychiatric disorders) | 0 (0) | 1 (1) | 1 (1)
Confusional state (Psychiatric disorders) | 0 (0) | 1 (1) | 1 (1)
Insomnia (Psychiatric disorders) | 2 (2) | 0 (0) | 2 (2)
Mood altered (Psychiatric disorders) | 1 (1) | 0 (0) | 1 (1)
Panic attack (Psychiatric disorders) | 0 (0) | 1 (1) | 1 (1)
Sleep disorder (Psychiatric disorders) | 0 (0) | 2 (2) | 2 (2)
Chronic kidney disease (Renal and urinary disorders) | 0 (0) | 1 (1) | 1 (1)
Dysuria (Renal and urinary disorders) | 0 (0) | 2 (2) | 2 (2)
Haematuria (Renal and urinary disorders) | 1 (1) | 2 (2) | 3 (3)
Urethral stenosis (Renal and urinary disorders) | 0 (0) | 1 (1) | 1 (1)
Gynaecomastia (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 1 (1)
Asthma (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 3 (3) | 6 (6)
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 4 (5) | 4 (5)
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (2) | 3 (3)
Increased upper airway secretion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 1 (1)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2) | 2 (2)
Orthopnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 1 (1)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 1 (1)
Sputum discoloured (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 1 (1)
Erythema (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (2) | 2 (2)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 1 (1)
Night sweats (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 1 (1)
Photosensitivity reaction (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 1 (1)
Pruritus (Skin and subcutaneous tissue disorders) | 1 (1) | 3 (4) | 4 (5)
Pruritus generalised (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 1 (1)
Rash (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1) | 2 (2)
Skin fissures (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 1 (1)
Skin irritation (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (2) | 2 (2)
Urticaria (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 1 (1)
Injection (Surgical and medical procedures) | 0 (0) | 1 (1) | 1 (1)
Deep vein thrombosis (Vascular disorders) | 0 (0) | 1 (1) | 1 (1)
Flushing (Vascular disorders) | 2 (2) | 9 (14) | 11 (16)
Haematoma (Vascular disorders) | 0 (0) | 1 (1) | 1 (1)
Hot flush (Vascular disorders) | 0 (0) | 2 (14) | 2 (14)
Hypertension (Vascular disorders) | 2 (2) | 9 (9) | 11 (11)
Peripheral venous disease (Vascular disorders) | 0 (0) | 1 (1) | 1 (1)
Venous thrombosis limb (Vascular disorders) | 1 (1) | 0 (0) | 1 (1)
Haemorrhoids (Gastrointestinal disorders) | 1 (1) | 1 (1) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2017-01-09): https://cdn.clinicaltrials.gov/large-docs/87/NCT02651987/Prot_001.pdf
  • Statistical Analysis Plan (2020-01-13): https://cdn.clinicaltrials.gov/large-docs/87/NCT02651987/SAP_000.pdf